CLINICAL TRIAL: NCT05406180
Title: Postmarketing Surveillance Study for Use of Quadrivalent Influenza Vaccine (VaxigripTetra Inj.) Administered Via the Intramuscular Route in Subjects Aged 3 Years Old and Above in the Republic of Korea
Brief Title: Postmarketing Surveillance Study for Quadrivalent Influenza Vaccine (VaxigripTetra Inj.) in Subjects Aged 3 Years Old and Above
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: GQM13
Record Dates: First submitted 2022-05-19; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: VaxigripTetra inj. — Suspension for injection in a pre-filled syringe Injection intramuscular
  Other Names: Quadrivalent influenza vaccine (split-virion, inactivated) - QIV

SUMMARY:
The objective is to describe the safety profile after 1 dose of VaxigripTetra inj. administered in subjects aged 3 years old and above under routine clinical practice.

The planned duration of each subject's participation in the study will be 21 to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 years and above on the day of enrollment
* For subjects aged 3 to 18 years: Informed consent form has been signed and dated by the parent or other legally acceptable representative.
* For subjects 19 years and above: Informed consent form has been signed and dated by the subject.
* Receipt of one dose of VaxigripTetra inj. (on the day of inclusion) as part of routine clinical practice according to the approved local product insert

Exclusion Criteria:

- Participation at the time of study enrollment (or in the 4 weeks preceding the enrollment) or planned participation during the present study period in a clinical study investigating a vaccine, drug, medical device, or medical procedure

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects aged 3 years old and above will be enrolled after receipt of one dose of VaxigripTetra inj. during a routine health care visit. Subjects will be enrolled on the day of vaccination and will be followed-up for one vaccination whatever their age at enrolment. Therefore, in case of the subjects under 9 years old (between 3 to 8 years of age), who may receive two doses depending on their previous influenza vaccination history, only one dose (either first or second vaccination) for each subject will be accounted for the study. The planned duration of each subject's participation in the study will be 21 to 28 days.
  Planned number of subjects: 670 subjects aged 3 years old and above Planned number of country: 1 (Republic of Korea) Planned number of sites: 10
Sampling Method: Non-Probability Sample
Enrollment: 675 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with solicited injection site or systemic reactions | Up to 7 days after vaccination
  Percentage of participants reporting
  * injection site reactions: pain, erythema, swelling, induration, ecchymosis
  * systemic reactions: fever, headache, malaise, myalgia, shivering
Number of participants with unsolicited adverse events | Up to Day 28
  Percentage of participants with unsolicited (spontaneously reported) injection site reactions occurring within 28 days after each injection and unsolicited systemic AEs between each injection and up to 28 days after the last injection
Number of participants with serious adverse events (SAEs) | Up to Day 28
  Percentage of participants with SAEs, including AESIs, throughout the study

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Site 009, Donghae-si, Gangwon-do
  - Site 011, Changwon
  - Site 012, Gwangju
  - Site 003, Gyeonggi-do
  - Site 005, Gyeonggi-do
  - Site 010, Gyeonggi-do
  - Site 004, Incheon
  - Site 007, Incheon
  - Site 008, Incheon
  - Site 002, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://www.vivli.org

REFERENCES:
- [Derived] Lim S, Li X, Syrkina O, Fournier M. Post-marketing Surveillance of a Quadrivalent Influenza Vaccine (Vaxigrip Tetra) in South Korea. Infect Dis Ther. 2022 Oct;11(5):2035-2043. doi: 10.1007/s40121-022-00685-x. Epub 2022 Sep 7. PMID 36070176